CLINICAL TRIAL: NCT06519721
Title: Safety and Efficacy Study of Lenvatinib Combined With VIC-1911 for the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Safety and Efficacy Study of Lenvatinib Combined With VIC-1911 for the Treatment of Advanced HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-LY2022-024-B
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1: Accelerated titration phase (Experimental): Plan to enroll 3 patients. First, enroll 1 patient, give the initial dose of VIC-1911 25mg BID, observe for 1 week, if there is no dose-limiting toxicity (DLT), increase to 50mg BID. At the same time, enroll another 2 patients, give VIC-1911 25mg BID, observe for 1 week, if no DLT, increase to 50mg BID. Observe for 2 weeks at a dose of 50mg, if no DLT occurs, continue to increase to 75mg BID, observe for 4 weeks. If no DLT occurs, continue to increase by 25mg doses, with an observation period of 4 weeks, until one case of dose-limiting toxicity or two cases of moderate toxicity occur during the titration process, then reduce to the previous dose, and determine it as the final dosing regimen.
  Interventions: Drug: Lenvatinib Combined with VIC-1911
- Phase 2: Expansion phase (Experimental): According to the final dosing regimen selected, enroll 12 patients and observe for 3 months.
  Interventions: Drug: Lenvatinib Combined with VIC-1911

INTERVENTIONS:
Drug: Lenvatinib Combined with VIC-1911 — Oral administration:
  Lenvatinib:
  Take the clinically normal dose: ≤60Kg body weight, 8mg/day; >60Kg body weight, 12mg/day;
  VIC-1911:
  Phase 1: Accelerated titration phase Plan to enroll 3 patients. First, enroll 1 patient, give the initial dose of VIC-1911 25mg BID, observe for 1 week, if there is no dose-limiting toxicity (DLT), increase to 50mg BID. At the same time, enroll another 2 patients, give VIC-1911 25mg BID, observe for 1 week, if no DLT, increase to 50mg BID. Observe for 2 weeks at a dose of 50mg, if no DLT occurs, continue to increase to 75mg BID, observe for 4 weeks. If no DLT occurs, continue to increase by 25mg doses, with an observation period of 4 weeks, until one case of dose-limiting toxicity or two cases of moderate toxicity occur during the titration process, then reduce to the previous dose, and determine it as the final dosing regimen.
  Phase 2: Expansion phase According to the final dosing regimen selected, enroll 12 patients and observe for 3 months.

SUMMARY:
This study is a single-arm, open-label trial to clarify the safety and efficacy of the combined treatment of lenvatinib and VIC-1911 in patients with advanced liver cancer.

DETAILED DESCRIPTION:
This study is a single-arm, open-label trial to clarify the safety and efficacy of the combined treatment of lenvatinib and VIC-1911 in patients with advanced liver cancer.

Purpose of the Study:

To observe and determine the safety and efficacy of lenvatinib combined with VIC-1911 in the treatment of patients with advanced liver cancer.

Sample Size:

According to the research plan, the administration of the study medication is divided into two stages, with 3 patients enrolled in the accelerated titration phase and 12 patients in the expansion phase.

Study Subjects:

Patients with advanced HCC

ELIGIBILITY:
Inclusion Criteria:

* Gender unrestricted, age 18-75 years;
* HCC conforms to AASLD or EASL clinical diagnostic standards;
* HCC Barcelona Clinic Liver Cancer (BCLC) staging is C, with at least one measurable tumor in the liver (longest diameter ≥1cm);
* Liver function Child-Pugh Class A or Class B with a score of 7;
* ECOG score of 0-1;
* Platelet count ≥60×10^9/L, PT time prolongation ≤6 seconds.

Exclusion Criteria:

* Irreversible coagulation dysfunction, with obvious bleeding tendency;
* Patients who need long-term anticoagulation or antiplatelet treatment and cannot stop medication;
* Patients with unstable or active ulcers, gastrointestinal bleeding;
* Patients with untreated heart disease or poorly controlled hypertension as judged by the researcher;
* Severe dysfunction of important organs, such as severe cardiopulmonary dysfunction;
* Patients with hepatic encephalopathy or refractory ascites requiring treatment;
* Human Immunodeficiency Virus (HIV) infection;
* Active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection (activity defined as viral load > 20000 IU/mL), or HBV, HCV positive patients who refuse to accept standardized antiviral treatment;
* Inability to swallow oral medication.
* Gastrointestinal diseases that may affect the absorption or tolerance of the study medication.
* History of corneal epithelial cysts or other causes of blurred vision, or medical abnormalities found in ophthalmic screening.
* Known allergy to VIC-1911 or its components.
* Within 4 weeks before the study, radiotherapy or interventional therapy for the disease under study was performed;
* Other concurrent antitumor treatments;
* The researcher assesses that the patient cannot or is unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Objective Response Rate (ORR) is defined as the proportion of patients experiencing a complete or partial response to a treatment

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Progression-Free Survival (PFS) is defined as the length of time during a study that a patient with a known cancer diagnosis does not experience disease worsening or death due to the disease.
Overall Survival (OS) | 2 years
  Overall Survival (OS) is defined as the percentage of patients in a study or a group of patients who are alive for a certain period of time after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No